CLINICAL TRIAL: NCT04517864
Title: A PHASE 2a, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY INVESTIGATING THE SAFETY OF RITLECITINIB (PF-06651600) IN ADULT PARTICIPANTS WITH ALOPECIA AREATA
Brief Title: PLACEBO-CONTROLLED SAFETY STUDY OF RITLECITINIB (PF-06651600) IN ADULTS WITH ALOPECIA AREATA
Acronym: Allegro2a
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For business reasons
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: B7981037; 2020-001509-21 (EudraCT Number)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Alopecia Areata
Keywords: alopecia totalis; alopecia universalis; hair loss; alopecia; JAK; ritlecitinib; PF-06651600; double-blind; placebo-controlled; phase 2a
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Alopecia | interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm: PF-06651600 (Experimental): ritlecitinib 200 milligram (mg) once per day (QD) (four 50 mg tablets) for 4 weeks then ritlecitinib 50 mg tablet QD through month 24. At Month 9, participants assigned to this treatment arm will also receive 3 tablets of placebo for 4 weeks to maintain the blind with the other arm. After month 24, participants switch to 50 mg capsules, 1 QD, up to month 60.
  Interventions: Drug: PF-06651600
- Control Arm (Placebo) followed by active therapy extension (Other): matching comparator: placebo QD (4 tablets x 4 weeks then 1 tablet x 8 months) then ritlecitinib 200 mg QD (four 50 mg tablets) for 4 weeks then ritlecitinib 50 mg tablet QD through month 24. After month 24, participants switch to 50 mg capsules, 1 QD, up to month 60.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06651600 — 50 mg tablet, dosed as 200 mg QD or 50 mg QD 50 mg capsule, dosed as 50 mg QD
  Other Names: ritlecitinib
  Arms: Treatment Arm: PF-06651600
Drug: Placebo — tablet, dosed as 4 tablets QD or 1 tablet QD
  Arms: Control Arm (Placebo) followed by active therapy extension

SUMMARY:
This is a global Phase 2a randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of ritlecitinib in adults aged 18 to ≤50 years of age with ≥25% scalp hair loss due to Alopecia Areata (AA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alopecia areata, including alopecia totalis and alopecia universalis.
* At least 25% hair loss due to alopecia areata
* Must have normal hearing and normal brainstem auditory evoked potentials (BAEPs)
* Must have a normal neurological exam; can have a stable unilateral median neuropathy or ulnar neuropathy
* Signed informed consent
* Stable regimen for other medications before and during the study

Exclusion Criteria:

* Other significant medical conditions
* Occupational or recreational noise exposure
* History of peripheral neuropathy or first degree relative with a hereditary peripheral neuropathy
* HbA1c > or = 7.5% at Screening
* Recurrent or disseminated Herpes Zoster
* Active or chronic infection; or infection requiring hospitalization or IV antimicrobials within 6 months
* Active or latent (insufficiently treated) Hepatitis
* Active or latent (insufficiently treated) TB
* Concomitant medications associated with peripheral neurologic or hearing loss
* Protocol specific laboratory abnormalities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (23):
  - Marvel Clinical Research 002, LLC, Huntington Beach, California
  - University of California, Irvine, Irvine, California
  - Skin Care Research, LLC, Boca Raton, Florida
  - Skin Care Research, LLC, Hollywood, Florida
  - Kendall Adkisson, MD - Intracoastal Dermatology, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Y&L Advance Health Care Inc., d/b/a Elite Clinical Research, Miami, Florida
  - BRCR Medical Center Inc, Miramar, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Orlando Dermatology & Skin Cancer Surgery Center, Oviedo, Florida
  - USF Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - NorthShore University HealthSystem Dermatology Clinic, Skokie, Illinois
  - Washington University School of Medicine-Dermatology, St Louis, Missouri
  - University of New Mexico Department of Dermatology, Albuquerque, New Mexico
  - University of New Mexico Clinical & Translational Sciences Center, Albuquerque, New Mexico
  - Stony Brook Dermatology, Stony Brook, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Tekton Research, Inc., Austin, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Summit Clinical Research, LLC, Franklin, Virginia
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Australia (3):
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
- Canada (4):
  - Lynderm Research Inc., Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Sima Recherche, Verdun, Quebec
  - Centre de Recherche Saint-Louis, Québec
- Poland (8):
  - Niepubliczny Zaklad Opieki Zdrowotnej Specjalistyczny Osrodek Dermatologiczny "DERMAL", Bialystok
  - Centrum Medyczne Angelius Provita, Katowice
  - AWP Klinika Dermatologii Pod Fortem Anna Wojas-Pelc, Krakow
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - RCMed Oddzial Warszawa, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Przychodnia przy ul. Lowieckiej, Wroclaw
  - Centrum Medyczne Matusiak, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] King B, Soung J, Tziotzios C, Rudnicka L, Joly P, Gooderham M, Sinclair R, Mesinkovska NA, Paul C, Gong Y, Anway SD, Tran H, Wolk R, Zwillich SH, Lejeune A. Integrated Safety Analysis of Ritlecitinib, an Oral JAK3/TEC Family Kinase Inhibitor, for the Treatment of Alopecia Areata from the ALLEGRO Clinical Trial Program. Am J Clin Dermatol. 2024 Mar;25(2):299-314. doi: 10.1007/s40257-024-00846-3. Epub 2024 Jan 23. PMID 38263353
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 131 participants were screened for this study; 71 participants were enrolled and randomized to double-blind treatment and treated. All enrolled participants received tablets until Month 24 and then all but 2 switched to capsules at the start of Extension Phase.
Groups:
- Ritlecitinib 200/50/50 mg QD: In the 9-Month Placebo-Controlled Phase, each participant received ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of ritlecitinib 50 mg QD during the remainder of this treatment phase. In the 15-Month Active Therapy Extension Phase, each participant received 1 tablet of ritlecitinib 50 mg QD and 3 tablets of placebo QD during the initial 4-week period, and then received 1 tablet of ritlecitinib 50 mg QD during the remainder of this phase.
- Placebo -> Ritlecitinib 200/50 mg QD: In the 9-month Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period, and received 1 tablet of Placebo QD during the remainder of this treatment phase. In the 15-month Active Therapy Extension Phase, each participant received ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and then received 1 tablet of ritlecitinib 50 mg QD during the remainder of this treatment phase.
- Ritlecitinib 50 mg QD: In the treatment period 3 (TP3), participants continued to receive ritlecitinib 50 mg QD during extension phase for 18 months and followed up for 4 weeks post completion or discontinuation of study intervention in the follow-up phase.
Period: Placebo-Controlled Phase
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD | Ritlecitinib 50 mg QD
Started | 36 | 35 | 0
Completed | 32 | 33 | 0
Not Completed | 4 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Period: Active Therapy Extension Phase
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD | Ritlecitinib 50 mg QD
Started | 32 | 33 | 0
Completed | 21 | 24 | 0
Not Completed | 11 | 9 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 8 | 0
Period: Extension Phase
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD | Ritlecitinib 50 mg QD
Started | 0 | 0 | 45
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 45
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Study Terminated By Sponsor | 0 | 0 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Approved Drug Available for Indication | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants taking at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (9.64) | 34.2 (8.95) | 34.7 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 26 | 28 | 54
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Baseline Percentage of Nerve Fibers With Axonal Swelling [Mean (Standard Deviation); unit: Percentage of Nerve Fibers] | 1.8 (2.48) | 1.8 (2.07) | 1.8 (2.27)
Baseline Intraepidermal Nerve Fiber Density (IENFD) [Mean (Standard Deviation); unit: fibers/mm] | 10.2 (3.81) | 11.0 (3.95) | 10.6 (3.87)
Baseline Severity of Alopecia Tool (SALT) Scores for Non-AT/AU Participants [Mean (Standard Deviation); unit: Units on a scale] — Baseline SALT score for non-alopecia totalis (AT)/alopecia universalis (AU) participants: SALT was a quantitative assessment of alopecia severity based on scalp terminal hair loss performed by an experienced and qualified rater. Score parameters utilized a visual aid showing the division of the scalp hair into 4 quadrants (back, top of scalp, and both sides), with each of 4 quadrants given an accurate determination of the % of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Higher SALT score represents greater amount of hair loss.
  Units on a scale | 59.6 (30.31) | 53.7 (24.18) | 56.9 (27.55)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in I-V Interwave Latency on Brainstem Auditory Evoked Potentials (BAEP) at a Stimulus Intensity of 80 Decibels (dB) From the Right Side at Month 9
Description: BAEP interwave I-V latency (in milliseconds) was the primary endpoint for this study. High-intensity stimulation (80dB) was used. Participants had BAEP evaluations performed at the same evaluation center, by the same audiology professional using the same equipment, during the study. Audiology and BAEP evaluations were done on the same day, with audiology assessment first. If they could not be done on the same day, assessments had to be within 7 days of each other. A central reader was used for BAEP to confirm that locally read BAEP waves were labelled appropriately and at their peak so that latency were accurate. Central reading also ensured consistency in BAEP interpretation.
Time Frame: Baseline, Month 9 (Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase)
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millisecond (ms)
Groups:
- Ritlecitinib 200/50 mg QD: In the 9-month Placebo-Controlled Phase, each participant received Ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of Ritlecitinib 50 mg QD during the remainder of this treatment phase.
- Placebo: In the 9-month Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period, and received 1 tablet of Placebo QD during the remainder of this treatment phase.
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 31 | 32
Millisecond (ms) | 0.011 [-0.043 to 0.065] | -0.010 [-0.063 to 0.043]
Statistical Analysis 1: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; Linear Mixed-effects Model: baseline, treatment group, visit and treatment group by visit interaction as fixed effects; participant as a random effect; Least Squares Mean Difference = 0.021, 95% CI 2-sided [-0.056 to 0.097], Standard Error of Mean 0.0382

2. Primary Outcome: Change From Baseline in I-V Interwave Latency on BAEP at a Stimulus Intensity of 80 dB From the Left Side at Month 9
Description: BAEP interwave I-V latency was the primary endpoint for this study. High-intensity stimulation (80dB) was used. Participants had BAEP evaluations performed at the same evaluation center, by the same audiology professional using the same equipment, during the study. Audiology and BAEP evaluations were done on the same day, with audiology assessment first. If they could not be done on the same day, assessments had to be within 7 days of each other. A central reader was used for BAEP to confirm that locally read BAEP waves were labelled appropriately and at their peak so that latency were accurate. Central reading also ensured consistency in BAEP interpretation.
Time Frame: as for outcome 1
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: ms
Groups:
- Ritlecitinib 200/50 mg QD: In the 9-month Placebo-Controlled Phase, each participant received Ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of Ritlecitinib 50 mg QD during the remainder of that study phase.
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 31 | 32
ms | 0.031 [-0.012 to 0.075] | 0.022 [-0.020 to 0.065]
Statistical Analysis 1: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.009, 95% CI 2-sided [-0.052 to 0.070], Standard Error of Mean 0.0307

3. Secondary Outcome: Change From Baseline in I-V Interwave Latency on BAEP at 80 dB From the Right Side at Month 6
Description: High-intensity stimulation (80dB) was used. Participants had BAEP evaluations performed at the same evaluation center, by the same audiology professional using the same equipment, during the study. Audiology and BAEP evaluations were done on the same day, with audiology assessment first. If they could not be done on the same day, assessments had to be within 7 days of each other. A central reader was used for BAEP to confirm that locally read BAEP waves were labelled appropriately and at their peak so that latency were accurate. Central reading also ensured consistency in BAEP interpretation.
Time Frame: Baseline, Month 6 (Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase)
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: millisecond (ms)
Groups:
- Placebo: In the 9-month Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period, and received 1 tablet of Placebo QD during the remainder of that study phase.
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 34 | 34
millisecond (ms) | -0.030 [-0.072 to 0.011] | -0.024 [-0.065 to 0.017]
Statistical Analysis 1: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.006, 95% CI 2-sided [-0.065 to 0.053], Standard Error of Mean 0.0297

4. Secondary Outcome: Change From Baseline in I-V Interwave Latency on BAEP at 80 dB From the Right Side at Month 9E and 15E
Description: as for outcome 3
Time Frame: Baseline, Months 9E and 15E (Month 9/15 in the Active Therapy Extension Phase). Baseline was defined as the last non-missing measurement obtained before the first dose in the Placebo-controlled Phase.
Population: Overall number of participants analyzed included all participants who received at least 1 dose of study intervention. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Groups:
- Ritlecitinib 200/50/50 mg QD: In the 9-Month Placebo-Controlled Phase, each participant received ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of ritlecitinib 50 mg QD during the remainder of this treatment phase. In the 15-month Active Therapy Extension Phase, each participant received 1 tablet of ritlecitinib 50 mg QD and 3 tablets of placebo QD during the initial 4-week period, and then received 1 tablet of ritlecitinib 50 mg QD during the remainder of this treatment phase.
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
millisecond (ms)
  Month 9E (Month 9 in the Active Therapy Extension Phase): number analyzed (Participants) | 25 | 30
  Month 9E (Month 9 in the Active Therapy Extension Phase) | 0.010 (0.1233) | -0.033 (0.2448)
  Month 15E (Month 15 in the Active Therapy Extension Phase): number analyzed (Participants) | 24 | 28
  Month 15E (Month 15 in the Active Therapy Extension Phase) | 0.051 (0.1188) | 0.034 (0.2224)

5. Secondary Outcome: Change From Baseline in I-V Interwave Latency on BAEP at 80 dB From the Left Side at Month 6
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: millisecond (ms)
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 34 | 34
millisecond (ms) | 0.021 [-0.011 to 0.054] | -0.020 [-0.053 to 0.012]
Statistical Analysis 1: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.042, 95% CI 2-sided [-0.005 to 0.088], Standard Error of Mean 0.0235

6. Secondary Outcome: Change From Baseline in I-V Interwave Latency on BAEP at 80 dB From the Left Side at Month 9E and 15E
Description: as for outcome 3
Time Frame: Baseline, Month 9E and 15E (Month 9/15 in the Active Therapy Extension Phase). Baseline was defined as the last non-missing measurement obtained before the first dose in the Placebo-controlled Phase.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
millisecond (ms)
  Month 9E (Month 9 in the Active Therapy Extension Phase): number analyzed (Participants) | 25 | 30
  Month 9E (Month 9 in the Active Therapy Extension Phase) | 0.006 (0.1109) | 0.056 (0.1694)
  Month 15E (Month 15 in the Active Therapy Extension Phase): number analyzed (Participants) | 24 | 28
  Month 15E (Month 15 in the Active Therapy Extension Phase) | 0.024 (0.1044) | 0.017 (0.2339)

7. Secondary Outcome: Change From Baseline in Percentage of Intraepidermal Nerve Fiber (IENF) With Axonal Swelling in Skin Punch Biopsies at Month 9
Description: The endpoint "axonal dystrophy" referred to the percentage of IENF with axonal swellings. Axonal swellings were evaluated in peripheral skin punch biopsies from the distal part of lower extremities. Axonal swellings were counted by axon. Any IENF with single or multiple swellings was counted as a single event, ie, a single axon with axonal swellings. For each participant, data were reported as the percentage of IENF with any number of swellings. IENF was assessed at Day 1 and Month 9. Participants who had entered the Active Therapy Extension Phase at Month 6 had a skin punch biopsy taken at Month 6 for IENF assessments instead of at Month 9. The skin biopsy was collected before the start of Active Therapy Extension Phase.
Time Frame: Baseline, Month 9 (Month 6 for the 2 participants who entered the Active Therapy Extension Phase at Month 6). Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase.
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Median (Inter-Quartile Range); unit: Percentage of Nerve Fibers
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 32 | 33
Percentage of Nerve Fibers | 0.0 [-0.5 to 2.5] | 0.0 [-2.0 to 1.0]

8. Secondary Outcome: Change From Baseline in Percentage of IENFs With Axonal Swelling in Skin Punch Biopsies at Month 15E
Description: The endpoint "axonal dystrophy" referred to the percentage of IENF with axonal swellings. Axonal swellings were evaluated in peripheral skin punch biopsies from the distal part of lower extremities. Axonal swellings were counted by axon. Any IENF with single or multiple swellings was counted as a single event, ie, a single axon with axonal swellings. For each participant, data were reported as the percentage of IENF with any number of swellings.
Time Frame: Baseline, Month 15E (Month 15 in the Active Therapy Extension Phase). Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percentage of Nerve Fibers
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
Percentage of Nerve Fibers | 0 [-1.0 to 0] | 0 [-1.0 to 0]

9. Secondary Outcome: Change From Baseline in Intraepidermal Nerve Fiber Density (IENFD) in Skin Punch Biopsies at Month 9
Description: IENFD was evaluated in peripheral skin punch biopsies from the distal part of lower extremities. IENFD was measured by counting the number of fibers and fiber branches that independently crossed the dermal-epidermal barrier (basement membrane). Secondary branching was excluded from quantification and fragments were not counted. The length of the histology section was measured (mm) and the linear epidermal nerve fiber density was reported as number of intraepidermal nerve fibers/mm.
Time Frame: as for outcome 7
Population: Analysis population included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 32 | 33
fibers/mm | -0.4 (3.90) | -0.2 (2.72)

10. Secondary Outcome: Change From Baseline in IENFD in Skin Punch Biopsies at Month 15E
Description: as for outcome 9
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
fibers/mm | 0.2 (2.85) | -1.1 (3.51)

11. Secondary Outcome: Change From Baseline in Amplitude of Wave V on BAEP at a Stimulus Intensity of 80 dB From the Right Side at Month 6 and Month 9
Description: High-intensity stimulation (80dB) was used. Participants had BAEP evaluations performed at the same evaluation center, by the same audiology professional using the same equipment, during the study. Audiology and BAEP evaluations were done on the same day, with audiology assessment first. If they could not be done on the same day, assessments had to be within 7 days of each other. A central reader was used for BAEP to confirm that locally read BAEP waves were labelled appropriately and at their peak so that amplitude data were accurate. Central reading also ensured consistency in BAEP interpretation.
Time Frame: Baseline, Month 6 and Month 9 (Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase)
Population: Analysis population included all participants who received at least 1 dose of study intervention. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Least Squares Mean (95% Confidence Interval); unit: Microvolts (μV)
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 34 | 34
Microvolts (μV)
  Month 6 | -0.031 [-0.063 to 0] | -0.017 [-0.048 to 0.015]
  Month 9: number analyzed (Participants) | 31 | 32
  Month 9 | -0.051 [-0.085 to -0.018] | 0.008 [-0.025 to 0.041]
Statistical Analysis 1: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Month 6; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.015, 95% CI 2-sided [-0.059 to 0.030], Standard Error of Mean 0.0224
Statistical Analysis 2: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Month 9; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.060, 95% CI 2-sided [-0.107 to -0.012], Standard Error of Mean 0.0236

12. Secondary Outcome: Change From Baseline in Amplitude of Wave V on BAEP at a Stimulus Intensity of 80 dB From the Right Side at Month 9E and 15E
Description: as for outcome 11
Time Frame: Baseline, Month 9E and 15E (Month 9 and 15 in the Active Therapy Extension Phase). Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
μV
  Month 9E (Month 9 in the Active Therapy Extension Phase): number analyzed (Participants) | 25 | 30
  Month 9E (Month 9 in the Active Therapy Extension Phase) | -0.052 (0.1109) | -0.025 (0.1649)
  Month 15E (Month 15 in the Active Therapy Extension Phase): number analyzed (Participants) | 24 | 28
  Month 15E (Month 15 in the Active Therapy Extension Phase) | -0.065 (0.1513) | -0.042 (0.1214)

13. Secondary Outcome: Change From Baseline in Amplitude of Wave V on BAEP at a Stimulus Intensity of 80 dB From the Left Side at Month 6 and Month 9
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: μV
Groups:
- Ritlecitinib 200/50 mg QD: In the Placebo-Controlled Phase, each participant received Ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of Ritlecitinib 50 mg QD during the remainder of that study phase.
- Placebo: In the Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period, and received 1 tablet of Placebo QD during the remainder of that study phase.
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 34 | 34
μV
  Month 6 | -0.047 [-0.082 to -0.013] | -0.019 [-0.053 to 0.015]
  Month 9: number analyzed (Participants) | 31 | 32
  Month 9 | -0.045 [-0.082 to -0.008] | -0.049 [-0.085 to -0.012]
Statistical Analysis 1: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Month 6; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.028, 95% CI 2-sided [-0.076 to 0.020], Standard Error of Mean 0.0242
Statistical Analysis 2: Comparison: Ritlecitinib 200/50 mg QD vs Placebo; Month 9; Test type: Superiority; Mixed Models Analysis — There was no formal statistical hypothesis testing for this study, and hence there was no P-value; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.003, 95% CI 2-sided [-0.049 to 0.056], Standard Error of Mean 0.0261

14. Secondary Outcome: Change From Baseline in Amplitude of Wave V on BAEP at a Stimulus Intensity of 80 dB From the Left Side at Month 9E and 15E
Description: as for outcome 11
Time Frame: as for outcome 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
μV
  Month 9E: number analyzed (Participants) | 25 | 30
  Month 9E | -0.058 (0.1209) | -0.025 (0.1307)
  Month 15E: number analyzed (Participants) | 24 | 28
  Month 15E | -0.047 (0.1314) | -0.023 (0.1217)

15. Secondary Outcome: Number of Participants With Absence of Wave V on BAEP at Stimulus Intensities Ranging From 80 dB to 40 dB From Right Side up to Month 9
Description: Absence of wave V on BAEP at stimulus intensities ranging from 80dB to 40dB were summarized descriptively using number of participants by treatment group at each intensity level.
  At Month 9, 1 participant in 200/50 mg had absence of Wave V on BAEP at a stimulus intensity of 40 dB on the right side. The event was unilateral and showed fluctuations in the presence or absence of Wave V at various intensities on repeat assessments starting at Month 6.
Time Frame: Baseline, Month 6 and 9 (Baseline was defined as the last non-missing measurement obtained before the first dose in the Placebo-Controlled Phase)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 36 | 35
Participants
  Baseline - 80 dB of normal hearing level (nHL) | 0 | 0
  Baseline - 70 dB nHL | 0 | 0
  Baseline - 60 dB nHL | 0 | 0
  Baseline - 50 dB nHL | 0 | 0
  Baseline - 40 dB nHL | 0 | 0
  Month 6 - 80 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 80 dB nHL | 0 | 0
  Month 6 - 70 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 70 dB nHL | 0 | 0
  Month 6 - 60 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 60 dB nHL | 0 | 0
  Month 6 - 50 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 50 dB nHL | 0 | 0
  Month 6 - 40 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 40 dB nHL | 0 | 0
  Month 9 - 80 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 80 dB nHL | 0 | 0
  Month 9 - 70 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 70 dB nHL | 0 | 0
  Month 9 - 60 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 60 dB nHL | 0 | 0
  Month 9 - 50 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 50 dB nHL | 0 | 0
  Month 9 - 40 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 40 dB nHL | 1 | 0

16. Secondary Outcome: Number of Participants With Absence of Wave V on BAEP at Stimulus Intensities Ranging From 80 dB to 40 dB From Right Side at Baseline, Month 3E, 6E, 9E and 15E
Description: Absence of wave V on BAEP at stimulus intensities ranging from 80dB to 40dB were summarized using number of participants by treatment group at each intensity level.
  All participants had Wave V on BAEP present at stimulus intensities ranging from 80 dB to 40 dB up to Month 15E except for 1 participant. At Month 9 (TP1), 1 participant in 200/50/50 mg had absence of Wave V on BAEP at a stimulus intensity of 40 dB on the right side. Fluctuations were seen in the presence or absence of Wave V at various intensities on repeat assessments starting at Month 6 on the right side.
Time Frame: Baseline, Month 3E, 6E, 9E and 15E (Baseline was defined as the last non-missing measurement obtained before the first dose in the Placebo-Controlled Phase)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
Participants
  Baseline - 80 dB nHL | 0 | 0
  Baseline - 70 dB nHL | 0 | 0
  Baseline - 60 dB nHL | 0 | 0
  Baseline - 50 dB nHL | 0 | 0
  Baseline - 40 dB nHL | 0 | 0
  Month 3E - 80 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 80 dB nHL | 0 | 0
  Month 3E - 70 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 70 dB nHL | 0 | 0
  Month 3E - 60 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 60 dB nHL | 0 | 0
  Month 3E - 50 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 50 dB nHL | 0 | 0
  Month 3E - 40 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 40 dB nHL | 0 | 0
  Month 6E - 80 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 80 dB nHL | 0 | 0
  Month 6E - 70 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 70 dB nHL | 0 | 0
  Month 6E - 60 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 60 dB nHL | 0 | 0
  Month 6E - 50 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 50 dB nHL | 0 | 0
  Month 6E - 40 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 40 dB nHL | 0 | 0
  Month 9E - 80 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 80 dB nHL | 0 | 0
  Month 9E - 70 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 70 dB nHL | 0 | 0
  Month 9E - 60 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 60 dB nHL | 0 | 0
  Month 9E - 50 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 50 dB nHL | 1 | 0
  Month 9E - 40 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 40 dB nHL | 1 | 0
  Month 15E - 80 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 80 dB nHL | 0 | 0
  Month 15E - 70 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 70 dB nHL | 0 | 0
  Month 15E - 60 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 60 dB nHL | 0 | 0
  Month 15E - 50 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 50 dB nHL | 0 | 0
  Month 15E - 40 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 40 dB nHL | 0 | 0

17. Secondary Outcome: Number of Participants With Absence of Wave V on BAEP at Stimulus Intensities Ranging From 80 dB to 40 dB From Left Side up to Month 9
Description: Absence of wave V on BAEP at stimulus intensities ranging from 80dB to 40dB were summarized descriptively using number of participants by treatment group at each intensity level.
Time Frame: as for outcome 15
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 36 | 35
Participants
  Baseline - 80 dB nHL | 0 | 0
  Baseline - 70 dB nHL | 0 | 0
  Baseline - 60 dB nHL | 0 | 0
  Baseline - 50 dB nHL | 0 | 0
  Baseline - 40 dB nHL | 0 | 0
  Month 6 - 80 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 80 dB nHL | 0 | 0
  Month 6 - 70 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 70 dB nHL | 0 | 0
  Month 6 - 60 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 60 dB nHL | 0 | 0
  Month 6 - 50 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 50 dB nHL | 0 | 0
  Month 6 - 40 dB nHL: number analyzed (Participants) | 34 | 34
  Month 6 - 40 dB nHL | 0 | 0
  Month 9 - 80 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 80 dB nHL | 0 | 0
  Month 9 - 70 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 70 dB nHL | 0 | 0
  Month 9 - 60 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 60 dB nHL | 0 | 0
  Month 9 - 50 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 50 dB nHL | 0 | 0
  Month 9 - 40 dB nHL: number analyzed (Participants) | 31 | 32
  Month 9 - 40 dB nHL | 0 | 0

18. Secondary Outcome: Number of Participants With Absence of Wave V on BAEP at Stimulus Intensities Ranging From 80 dB to 40 dB From Left Side at Baseline, Month 3E, 6E, 9E and 15E
Description: Absence of wave V on BAEP at stimulus intensities ranging from 80dB to 40dB were summarized descriptively using number of participants by treatment group at each intensity level.
  All participants had Wave V on BAEP present at stimulus intensities ranging from 80 dB to 40 dB up to Month 15E except for 1 participant. At Month 9 (TP1), 1 participant in 200/50/50 mg had absence of Wave V on BAEP at a stimulus intensity of 40 dB on the right side. Fluctuations were seen in the presence or absence of Wave V at various intensities on repeat assessments starting at Month 6 on the right side.
Time Frame: as for outcome 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
Participants
  Baseline - 80 dB nHL | 0 | 0
  Baseline - 70 dB nHL | 0 | 0
  Baseline - 60 dB nHL | 0 | 0
  Baseline - 50 dB nHL | 0 | 0
  Baseline - 40 dB nHL | 0 | 0
  Month 3E - 80 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 80 dB nHL | 0 | 0
  Month 3E - 70 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 70 dB nHL | 0 | 0
  Month 3E - 60 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 60 dB nHL | 0 | 0
  Month 3E - 50 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 50 dB nHL | 0 | 0
  Month 3E - 40 dB nHL: number analyzed (Participants) | 1 | 0
  Month 3E - 40 dB nHL | 0 | 0
  Month 6E - 80 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 80 dB nHL | 0 | 0
  Month 6E - 70 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 70 dB nHL | 0 | 0
  Month 6E - 60 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 60 dB nHL | 0 | 0
  Month 6E - 50 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 50 dB nHL | 0 | 0
  Month 6E - 40 dB nHL: number analyzed (Participants) | 1 | 1
  Month 6E - 40 dB nHL | 0 | 0
  Month 9E - 80 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 80 dB nHL | 0 | 0
  Month 9E - 70 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 70 dB nHL | 0 | 0
  Month 9E - 60 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 60 dB nHL | 0 | 0
  Month 9E - 50 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 50 dB nHL | 0 | 0
  Month 9E - 40 dB nHL: number analyzed (Participants) | 25 | 30
  Month 9E - 40 dB nHL | 0 | 0
  Month 15E - 80 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 80 dB nHL | 0 | 0
  Month 15E - 70 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 70 dB nHL | 0 | 0
  Month 15E - 60 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 60 dB nHL | 0 | 0
  Month 15E - 50 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 50 dB nHL | 0 | 0
  Month 15E - 40 dB nHL: number analyzed (Participants) | 24 | 28
  Month 15E - 40 dB nHL | 0 | 0

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Seriousness of an AE was assessed under the criteria of serious adverse event (SAE). An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect, etc. Treatment-emergent events were with onset date occurring during the on-treatment period. Relatedness to study treatment was determined by the investigator.
Time Frame: Approximately 16 months
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase: In the 9-month Placebo-Controlled Phase, each participant received Ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of Ritlecitinib 50 mg QD during the remainder of this treatment phase.
- Placebo - Placebo-Controlled Phase: In the 9-month Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period, and received 1 tablet of Placebo QD during the remainder of this treatment phase.
- Ritlecitinib 50 mg QD - Active Therapy Extension Phase: In the 15-month Active Therapy Extension Phase, each participant received 1 tablet QD of Ritlecitinib 50 mg and 3 tablets of placebo QD during the initial 4-week period, and then received 1 tablet of Ritlecitinib 50 mg QD during the remainder of this phase.
- Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase: In the 15-month Active Therapy Extension Phase, each participant received Ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and then received 1 tablet of Ritlecitinib 50 mg QD during the remainder of this phase.
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase
Number analyzed (Participants) | 36 | 35 | 32 | 31
Participants
  TEAE (All-Causality) | 29 | 22 | 3 | 3
  TEAE (Treatment-Related) | 9 | 5 | 0 | 1
  TESAE (All-Causality) | 0 | 1 | 1 | 0
  TESAE (Treatment-Related) | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants Who Discontinued From Study Due to Adverse Event (AEs)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Participants who had an AE record that indicated that the AE caused the participant to be discontinued from the study. Relatedness to study treatment was determined by the investigator.
Time Frame: Approximately 16 months
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Placebo-Controlled Phase: In the 9-month Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period and received 1 tablet of Placebo QD during the remainder of this treatment phase.
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase
Number analyzed (Participants) | 36 | 35 | 32 | 31
Participants
  Due to All-Causality AEs | 0 | 0 | 1 | 0
  Due to Treatment-Related AEs | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to AE and Continued Study
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. This Outcome Measures presented the number of participants who had an AE record that indicated that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study. Relatedness to study treatment was determined by the investigator.
Time Frame: Approximately 16 months
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase: In the 9-month Placebo-Controlled Phase, each participant received Ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and received 1 tablet of Ritlecitinib 50 mg QD during the remainder of that study phase.
- Placebo - Placebo-Controlled Phase: In the 9-month Placebo-Controlled Phase, each participant received a total of 4 tablets of Placebo QD during the initial 4-week period, and received 1 tablet of Placebo QD during the remainder of that study phase.
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase
Number analyzed (Participants) | 36 | 35 | 32 | 31
Participants
  Due to All-Causality AEs | 1 | 0 | 0 | 0
  Due to Treatment-Related AEs | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Temporary Drug Discontinuation Due to AEs
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with temporary drug discontinuation due to both all-causality and treatment-related AEs are presented below. Relatedness to study treatment was determined by the investigator.
Time Frame: Approximately 16 months
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase
Number analyzed (Participants) | 36 | 35 | 32 | 31
Participants
  Due to All-Causality AEs | 6 | 1 | 0 | 0
  Due to Treatment-Related AEs | 3 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Oral, tympanic, or axillary temperature, pulse rate, respiratory rate, and blood pressure (BP) were assessed. BP and pulse measurements were assessed in a chair, back supported and arms bared (free of restrictions such as rolled-up sleeves, etc) and supported at heart level. Measurements were taken on the same arm at each visit (preferably non-dominant) with a completely automated device. Pulse rate was measured at approximately the same time as BP for a minimum of 30 seconds. BP and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (eg, television, cell phones). Participants refrained from smoking or ingesting caffeine during the 30 minutes preceding the measurements. The clinical significance was determined by the investigator.
Time Frame: Approximately 16 months
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase
Number analyzed (Participants) | 36 | 35 | 32 | 31
Participants | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values
Description: Safety laboratory assessments included the categories of Hematology, Chemistry, Urinalysis and other tests. The clinical significance was determined by the investigator.
Time Frame: Approximately 16 months
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase
Number analyzed (Participants) | 36 | 35 | 32 | 31
Participants | 0 | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in Overall Severity of Alopecia Tool (SALT) Scores up to Month 9
Description: SALT is a quantitative assessment of AA severity based on scalp terminal hair loss. The overall SALT score included hair loss regardless of etiology (ie, scalp hair loss due to both non-AA and AA) and was collected at study visits. The Overall SALT Score ranged from 0 to 100%, with higher scores representing greater amount of hair loss.
Time Frame: Baseline, Months 3, 6 and 9 (Baseline was defined as the last non-missing measurement obtained before the first dose in the placebo-controlled phase)
Population: Analysis population included all randomized participants taking at least 1 dose of study intervention. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 35 | 35
Units on a scale
  Month 3 | -23.0 [-29.70 to -16.25] | -2.7 [-9.39 to 4.06]
  Month 6: number analyzed (Participants) | 34 | 35
  Month 6 | -35.2 [-44.55 to -25.81] | -5.1 [-14.44 to 4.18]
  Month 9: number analyzed (Participants) | 32 | 31
  Month 9 | -38.2 [-47.46 to -28.86] | -6.8 [-16.08 to 2.40]

26. Secondary Outcome: Change From Baseline in Overall SALT Scores at Month 3E, 6E, 9E, 12E and 15E
Description: as for outcome 25
Time Frame: Baseline, Month 3E, 6E, 9E, 12E and 15E (Month 3, 6, 9, 12 and 15 in the Active Therapy Extension Phase). Baseline was defined as the last non-missing measurement obtained before the first dose in the Placebo-Controlled Phase.
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
Units on a scale
  Baseline | 69.7 (31.56) | 69.6 (29.59)
  Change at Month 3E: number analyzed (Participants) | 32 | 33
  Change at Month 3E | -41.7 (33.98) | -38.7 (33.49)
  Change at Month 6E: number analyzed (Participants) | 29 | 30
  Change at Month 6E | -38.0 (29.88) | -43.4 (34.13)
  Change at Month 9E: number analyzed (Participants) | 26 | 30
  Change at Month 9E | -38.7 (29.90) | -46.6 (34.14)
  Change at Month 12E: number analyzed (Participants) | 25 | 29
  Change at Month 12E | -41.6 (29.67) | -48.9 (34.77)
  Change at Month 15E: number analyzed (Participants) | 24 | 28
  Change at Month 15E | -44.6 (28.51) | -49.9 (34.40)

27. Secondary Outcome: Change From Baseline in Alopecia Areata - Severity of Alopecia Tool (AA-SALT) Score up to Month 9
Description: SALT is a quantitative assessment of AA severity based on scalp terminal hair loss. AA-SALT is the amount of scalp hair loss due to AA. AA SALT score in Placebo-Controlled Phase = overall SALT score - non-AA SALT score (The non-AA SALT score only took into account scalp hair loss other than that due to AA and was required to be assessed only at Month 9 [or Month 6 for those who entered the Active Therapy Extension Phase at Month 6] in Placebo-Controlled Phase). The AA-SALT Score ranged from 0 to 100%, with higher scores representing greater amount of hair loss.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 35 | 35
Units on a scale
  Month 3 | -23.0 [-29.70 to -16.25] | -2.7 [-9.39 to 4.06]
  Month 6: number analyzed (Participants) | 34 | 35
  Month 6 | -35.2 [-44.55 to -25.81] | -5.1 [-14.44 to 4.18]
  Month 9: number analyzed (Participants) | 32 | 31
  Month 9 | -38.2 [-47.46 to -28.87] | -6.8 [-16.08 to 2.40]

28. Secondary Outcome: Change From Baseline in AA-SALT Score at Month 3E, 6E, 9E, 12E and 15E
Description: SALT is a quantitative assessment of AA severity based on scalp terminal hair loss. AA-SALT is the amount of scalp hair loss due to AA. AA SALT score = overall SALT score - non-AA SALT score (The non-AA SALT score only took into account scalp hair loss other than that due to AA and was required to be assessed only at Month 9 [or Month 6 for those who entered the Active Therapy Extension Phase at Month 6] in Placebo-Controlled Phase). The AA-SALT Score ranged from 0 to 100%, with higher scores representing greater amount of hair loss.
Time Frame: Baseline, Month 3E, 6E, 9E, 12E and 15E (Baseline was defined as the last non-missing measurement obtained before the first dose in the Placebo-Controlled Phase)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
Units on a scale
  Baseline | 67.0 (33.52) | 69.5 (29.67)
  Change at Month 3E: number analyzed (Participants) | 32 | 33
  Change at Month 3E | -41.7 (33.97) | -39.4 (32.89)
  Change at Month 6E: number analyzed (Participants) | 29 | 30
  Change at Month 6E | -38.0 (29.87) | -44.2 (33.37)
  Change at Month 9E: number analyzed (Participants) | 26 | 30
  Change at Month 9E | -38.7 (29.90) | -47.4 (33.36)
  Change at Month 12E: number analyzed (Participants) | 25 | 29
  Change at Month 12E | -41.6 (29.70) | -49.7 (33.92)
  Change at Month 15E: number analyzed (Participants) | 24 | 28
  Change at Month 15E | -44.8 (28.37) | -50.8 (33.49)

29. Secondary Outcome: Number of Participants With Patient's Global Impression of Change (PGI-C) Response up to Month 9
Description: The PGI-C asked the participants to evaluate the improvement or worsening of their AA as compared to the start of the study using a single item, "Since the start of the study, my alopecia areata has: …". The participants selected one of seven responses ranging from "greatly improved" to "greatly worsened". This Outcome Measure presented the number of participants with PGI-C response which was defined as "greatly improved" or "moderately improved". Participants with missing PGI-C scores were considered as non-responders.
Time Frame: Months 1, 3, 6 and 9
Population: Analysis population included all randomized participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50 mg QD | Placebo
Number analyzed (Participants) | 36 | 35
Participants
  Month 1 | 4 | 3
  Month 3 | 20 | 6
  Month 6 | 21 | 10
  Month 9 | 19 | 6

30. Secondary Outcome: Number of Participants With PGI-C Response at 3E, 6E, 9E, 12E and 15E
Description: as for outcome 29
Time Frame: Month 3E, 6E, 9E, 12E and 15E
Population: Analysis population included all randomized participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 200/50/50 mg QD | Placebo -> Ritlecitinib 200/50 mg QD
Number analyzed (Participants) | 36 | 35
Participants
  Month 3E | 22 | 22
  Month 6E | 16 | 20
  Month 9E | 20 | 18
  Month 12E | 17 | 18
  Month 15E | 17 | 18

31. Secondary Outcome: Number of Participants With TEAEs and TESAEs: Extension Phase (TP3)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Seriousness of an AE was assessed under the criteria of SAE. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect, etc. Treatment-emergent events were with onset date occurring during the on-treatment period. Relatedness to study treatment was determined by the investigator.
Time Frame: From first dose of treatment up to 28 days follow up after last dose of study treatment (Approximately 19 months)
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 50 mg QD
Number analyzed (Participants) | 45
Participants
  TEAEs | 19
  TESAEs | 1

32. Secondary Outcome: Number of Participants Who Discontinued From Study Due to AEs: Extension Phase (TP3)
Description: as for outcome 20
Time Frame: From first dose of treatment up to 28 days follow up after last dose of study treatment (Approximately 19 months)
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 50 mg QD
Number analyzed (Participants) | 45
Participants | 1

33. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to AE and Continued Study: Extension Phase (TP3)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. This outcome measure presented the number of participants who had an AE record that indicated that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study. Relatedness to study treatment was determined by the investigator.
Time Frame: From first dose of treatment up to 28 days follow up after last dose of study treatment (Approximately 19 months)
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 50 mg QD
Number analyzed (Participants) | 45
Participants | 0

34. Secondary Outcome: Number of Participants With Temporary Drug Discontinuation Due to AEs: Extension Phase (TP3)
Description: as for outcome 22
Time Frame: From first dose of treatment up to 28 days follow up after last dose of study treatment (Approximately 19 months)
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 50 mg QD
Number analyzed (Participants) | 45
Participants | 1

35. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs: Extension Phase (TP3)
Description: Oral, tympanic, or axillary temperature, pulse rate, respiratory rate, and blood pressure (BP) were assessed. BP and pulse measurements were assessed in a chair, back supported and arms bared (free of restrictions such as rolled-up sleeves, etc) and supported at heart level. Measurements were taken on the same arm at each visit (preferably non-dominant) with a completely automated device. Pulse rate was measured at approximately the same time as BP for a minimum of 30 seconds. BP and pulse measurements preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (eg, television, cell phones). Participants were refrained from smoking or ingesting caffeine during the 30 minutes preceding the measurements. The clinical significance was determined by the investigator.
Time Frame: From screening up to 28 days follow up after last dose of study treatment (maximum up to 19 months)
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 50 mg QD
Number analyzed (Participants) | 45
Participants | 0

36. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values: Extension Phase (TP3)
Description: as for outcome 24
Time Frame: From screening up to 28 days after last dose of study treatment (maximum up to 19 months)
Population: Analysis population included all participants taking at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 50 mg QD
Number analyzed (Participants) | 45
Participants | 0

ADVERSE EVENTS:
Time Frame: Placebo controlled phase (TP1) & Active therapy extension phase (TP2): 24 months, Extension phase (TP3): From first dose of treatment up to 28 days follow up after last dose of study treatment (Approximately 19 months)
Description: Same event may appear as both an AE and SAE.However,what is presented are distinct events.Event may be categorized as serious in 1 participant,as non-serious in another participant,or 1 participant may have experienced both serious and non-serious event during study.Analysis population=all participants taking at least 1dose of study intervention.
Groups:
- Ritlecitinib 50 mg QD - Active Therapy Extension Phase: In the 15-month Active Therapy Extension Phase, each participant received 1 tablet of ritlecitinib 50 mg QD and 3 tablets of placebo QD during the initial 4-week period, and then received 1 tablet of ritlecitinib 50 mg QD during the remainder of this treatment phase.
- Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase: In the 15-month Active Therapy Extension Phase, each participant received ritlecitinib 200 mg QD (50 mg/tablet ×4) during the initial 4-week period, and then received 1 tablet of ritlecitinib 50 mg QD during the remainder of this treatment phase.
- Ritlecitinib 50 mg QD: Extension Phase: In the treatment period 3 (TP3), participants continued to receive ritlecitinib 50 mg QD during extension phase for 18 months and followed up for 4 weeks post completion or discontinuation of study intervention in the follow-up phase.
Arm/Group | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase | Placebo - Placebo-Controlled Phase | Ritlecitinib 50 mg QD - Active Therapy Extension Phase | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase | Ritlecitinib 50 mg QD: Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35 | 0/32 | 0/33 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/35 | 2/32 | 1/33 | 1/45
Other Adverse Events (participants affected / at risk) | 23/36 | 17/35 | 16/32 | 12/33 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase (N=36) | Placebo - Placebo-Controlled Phase (N=35) | Ritlecitinib 50 mg QD - Active Therapy Extension Phase (N=32) | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase (N=33) | Ritlecitinib 50 mg QD: Extension Phase (N=45)
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Takayasu's arteritis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 was used for Ritlecitinib 200/50/50 mg QD and Placebo -> Ritlecitinib 200/50 mg QD Cohort. MedDRA v27.0 was used for Ritlecitinib 50 mg QD: Extension Phase Cohort.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritlecitinib 200/50 mg QD - Placebo-Controlled Phase (N=36) | Placebo - Placebo-Controlled Phase (N=35) | Ritlecitinib 50 mg QD - Active Therapy Extension Phase (N=32) | Ritlecitinib 200/50 mg QD - Active Therapy Extension Phase (N=33) | Ritlecitinib 50 mg QD: Extension Phase (N=45)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0
Acne pustular (Infections and infestations) | 4 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 3 | 5 | 6 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 2 | 2
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 0 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT04517864/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT04517864/SAP_003.pdf